CLINICAL TRIAL: NCT01415843
Title: Do Implicit and Explicit Learning Strategies Applied During Gait Re-education Influence Concurrent Expression of Associated Reactions in Individuals With Hemiplegia? Phase 1a
Brief Title: Observation of Physiotherapy Treatment Sessions - Exploring What Happens in Physiotherapy for Patients After Stroke.
Status: Completed | Type: Observational
Sponsor: University of Southampton (Other)
Responsible Party: Sponsor
Other Study IDs: 09/H0504/80
Record Dates: First submitted 2011-08-11; First posted 2011-08-12 (Estimated); Last update posted 2021-04-20 (Actual); Status verified 2021-04

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is the first phase of a study that will investigate the effects that different approaches to physiotherapy have on the expression of associated reactions. During this phase, current practice among neuro-physiotherapists will be explored in relation to: the learning strategies used in stroke rehabilitation, the common interventions used in gait re-education, and the strategies adopted for the assessment and management of associated reactions.

DETAILED DESCRIPTION:
Associated reactions are unintended and involuntary arm movements, normally seen as bending of the wrist and elbow, that may occur after stroke when a person is doing something effortful such as walking.

The objectives are:

* To provide an insight into the learning strategies used by physiotherapists during the re-education of walking, including the verbal dialogue that takes place and any preferences (overt or subconscious) adopted for one type of learning strategy.
* To develop and refine a description of what is meant by the term "gait re-education"
* To provide an insight into how therapists currently manage associated reactions

This phase of the study will explore these objectives using direct non-participation observation of a number of physiotherapy treatment sessions. This will provide an insight into the nature of the therapy that takes place for retraining walking(e.g. the types of exercises commonly used) and the nature of the learning strategies frequently adopted, including the amount and content of explicit verbal instruction and feedback that is provided to patients.

ELIGIBILITY:
* has suffered a stroke
* is currently receiving active rehabilitation that includes gait re-education
* is exhibiting upper limb deficits
* is able to provide informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with stroke will be recruited from two NHS Trusts - Royal Bournemouth and Christchuch Hospitals NHS Foundation Trust and Southampton City Primary Care Trust.
Sampling Method: Non-Probability Sample
Enrollment: 8 (Actual)
Dates: Start 2010-01 (Actual); Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jane Burridge, Professor, Study Chair — University of Southampton
Locations (2):
- United Kingdom (2):
  - Royal Bournemouth and Christchurch NHS Foundation Trust, Bournemouth, Dorset
  - Southampton City Primary Care Trust, Southampton, Hampshire

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Johnson L, Burridge JH, Demain SH. Internal and external focus of attention during gait re-education: an observational study of physical therapist practice in stroke rehabilitation. Phys Ther. 2013 Jul;93(7):957-66. doi: 10.2522/ptj.20120300. Epub 2013 Apr 4. PMID 23559523